CLINICAL TRIAL: NCT02725463
Title: First-in-Human Early Feasibility Study of Safety, Tolerability and Efficacy for a Multichannel Vestibular Implant in Individuals With Bilateral Severe-to-Profound Loss of Vestibular Sensation
Brief Title: Multichannel Vestibular Implant Early Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Labyrinth Devices, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NA_00051349; R01DC013536 (NIH); JHU80640 (Other: Labyrinth Devices, LLC); 1U01DC019364 (NIH)
Record Dates: First submitted 2016-01-12; First posted 2016-04-01 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Other Disorders of Vestibular Function, Bilateral; Bilateral Vestibular Deficiency (BVD); Gentamicin Ototoxicity; Labyrinth Diseases; Vestibular Diseases; Sensation Disorders
Keywords: vestibular; implant; prosthesis; labyrinth; ototoxicity; gentamicin; oscillopsia; disequilibrium; dizziness; vestibulopathy; inner ear
MeSH Terms: conditions — Bilateral Vestibulopathy; Labyrinth Diseases; Vestibular Diseases; Sensation Disorders; Ototoxicity; Dysequilibrium syndrome; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vestibular implant (Experimental): Up to 30 participants will undergo implantation, activation and deactivation of a Labyrinth Devices MVI™ Multichannel Vestibular Implant System
  Interventions: Device: Labyrinth Devices MVI™ Multichannel Vestibular Implant

INTERVENTIONS:
Device: Labyrinth Devices MVI™ Multichannel Vestibular Implant

SUMMARY:
Although cochlear implants can restore hearing to individuals who have lost cochlear hair cell function, there is no adequately effective treatment for individuals suffering chronic imbalance, postural instability and unsteady vision due to loss of vestibular hair cell function. Preclinical studies have demonstrated that electrical stimulation of the vestibular nerve via a chronically implanted multichannel vestibular prosthesis can partially restore vestibular reflexes that maintain steady posture and vision. This pilot clinical feasibility study of a multichannel vestibular implant system will evaluate this approach in up to ten human subjects with bilateral vestibular deficiency due to gentamicin ototoxicity or other causes of inner ear dysfunction.

DETAILED DESCRIPTION:
The system used in this study is the (MVI)™ Multichannel Vestibular Implant System produced by Labyrinth Devices, LLC. It is similar to commercially available cochlear implants in that it includes an implanted stimulator powered and controlled by an external unit, which communicate with the implant across the skin via an inductive link. Unlike a cochlear implant, the implanted stimulator's electrode array is designed for implantation near the ends of the vestibular nerve. The implanted stimulator also includes additional magnets to help facilitate retention of the external unit on the scalp over the implant. The external unit includes a head-worn unit (for sensing head motion and delivering power and signals to the implanted stimulator) and a power and control unit containing a battery and microprocessor. Participants in this trial who meet candidacy criteria and who choose to proceed with implantation surgery, device activation and device deactivation will be asked to participate in a series of post-operative monitoring visits over a ≥1 year period.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 22.0-90 with bilateral vestibular deficiency not responsive to vestibular rehabilitation as determined by pre-inclusion history, vestibular testing and clinical examination
2. Hearing status: (1) Hearing in the candidate ear for implantation is equivalent to or worse than that in the contralateral ear; and (2) hearing in the contralateral ear is good enough to allow functional communication in case hearing in the implanted ear is lost after implantation. Specifically, the contralateral ear must satisfy all of the following criteria:

   1. 0.5/1/2/4 kHz pure-tone-average threshold (PTA) hearing better than (i.e., less than) 70 dB HL; and
   2. ear-specific sentence recognition score using the recorded AzBio Sentence Test presented at 60 dB SPL-A in quiet must be >60% when tested under either the unaided condition or, if 0.5/1/2/4 kHz PTA>50 dB, the best-aided condition; and
   3. ear-specific word recognition score using the recorded Consonant-Nucleus-Consonant (CNC) Word Recognition Test presented at 60 dBHL in quiet must be >60% when tested under either the unaided condition or, if 0.5/1/2/4 kHz PTA>50 dB, the best-aided condition
3. Caloric responses consistent with severe or profound bilateral loss of labyrinthine function, as indicated by one or more of the following: (a) summed speed of caloric responses to warm and cool supine caloric stimuli totaling <10°/sec per ear for each of both ears; (b) summed speed of ice water caloric responses during supine and prone head orientation tests totaling <10°/sec per ear for each of both ears; or (c) speed of ice water caloric responses during supine head orientation tests <5°/sec per ear for each of both ears, with a lack of nystagmus reversal on quickly flipping from supine to prone
4. Prior MRI imaging of the brain, internal auditory canals and cerebellopontine (CP) angle showing a patent labyrinth, present vestibular nerve, patent cochlea, present cochlear nerve, and absence of internal auditory canal/cerebellopontine angle tumors or other central causes of vestibulo-ocular reflex dysfunction or sensorineural hearing loss
5. Prior CT imaging of the temporal bones showing a facial nerve canal with normal caliber and course, middle ear without evidence of chronic otitis media or tympani membrane perforation or cholesteatoma, a mastoid cavity with adequate aeration for surgical access to each semicircular canal, skull thickness ≥3 mm at the planned well site, and scalp soft tissue thickness ≤7 mm. This criterion may be satisfied without additional imaging if an existing head CT or MRI already demonstrates those findings
6. Vaccinations as recommended per Johns Hopkins Listening Center protocols to reduce the risk of meningitis in subjects undergoing cochlear implantation, as described at this site: http://www.hopkinsmedicine.org/otolaryngology/specialty_areas/listencenter/vaccine.html
7. Motivated to travel to the study center, to undergo testing and examinations required for the investigational study, and to participate actively in a vestibular rehabilitation exercise regimen
8. The participant must agree not to swim or to use or operate vehicles, heavy machinery, powered tools or other devices that could pose a threat to the participant, to others, or to property throughout the duration of participation in the study and until at least 1 month after final deactivation of the MVI Implant

Exclusion Criteria:

1. Inability to understand the procedures and the potential risks involved as determined by study staff
2. Inability to participate in study procedures due to blindness, ≤ ±10° neck range of motion, cervical spine instability, ear canal stenosis or malformation sufficient to prevent caloric testing
3. Diagnosis of acoustic neuroma/vestibular schwannoma, chronic middle ear disease, cholesteatoma, or central nervous system causes of vestibulo-ocular reflex dysfunction, including chronic and continuing use of medications, drugs or alcohol at doses sufficiently great to interfere with vestibular compensation
4. Vestibular dysfunction known to be caused by reasons other than labyrinthine injury due to ototoxicity, ischemia, trauma, infection, Meniere's disease, or genetic defects known to act on hair cells
5. Lack of labyrinth patency or vestibular nerve as determined by MRI of the brain with attention to the internal acoustic meatus
6. Any contraindication to the planned surgery, anesthesia, device activation and deactivation, or participation in study assessments, as determined by the surgeon, anesthesiologist, or designee, including known intolerance of any materials used in any component of the investigational devices that will come in contact with the subject
7. History of myocardial infarction, coronary bypass surgery, or any percutaneous coronary intervention (PCI) within 6 months prior to screening
8. Orthopedic, neurologic or other nonvestibular pathologic conditions of sufficient severity to confound posture and gait testing or other tests used in the study to assay vestibular function.
9. Subjects with estimated glomerular filtration rate (GFR) < 30 ml/min (MDRD formula) at screening
10. Subjects with heart failure NYHA class III or IV
11. Subjects with Child-Pugh class C cirrhosis
12. A psychiatric disease or substance abuse history likely to interfere with protocol compliance
13. Contraindications to scleral coil eye movement testing, including monocular blindness and a history of fainting vagal reactions to prior eye manipulations would exclude subjects from eye coil testing
14. Inability to tolerate baseline testing protocols
15. Recent corneal injury
16. A history of cervical spine disease preventing head rotation
17. A history of fainting or vagal reactions prior to eye manipulations that would preclude 3D eye movement coil testing
18. Pregnancy, positive urine or serum pregnancy test at any time during study participation,
19. Ability to become pregnant combined with failure or refusal to consistently use a highly effective method of contraception from at least 1 month prior to implantation to not before 1 month after both device deactivation and conclusion of study participation. Highly effective contraception methods include:

    Total abstinence. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception for purposes of defining exclusion criteria for this study

    Female sterilization (surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before entering the study. A woman who has undergone oophorectomy without hysterectomy may participate in the study only after her reproductive status has been confirmed by subsequent hormone level assessment

    For female subjects of child-bearing potential, study participation is not excluded if the study candidate's male partner is the sole partner of the study candidate and has been vasectomized.

    Combination of any two of the following:

    Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example, hormone vaginal ring or transdermal hormone contraception

    Placement of an intrauterine device (IUD) or intrauterine system (IUS)

    Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository In case of use of oral contraception, women should have been stabile on the same pill for a minimum of 3 months before taking study treatment.
20. Women who are nursing/lactating
21. Any medical condition, judged by the investigator team, that is likely to interfere with a study candidate's participation in the study or likely to cause serious adverse events during the study.

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Identified adverse events to assess the safety and tolerability of the Labyrinth Devices Multichannel Vestibular Implant (MVI™) | Through study completion, an average of 1 year, that is: in visits 0 through 10
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events v4.3 (CTCAE v4.3)
Assess the feasibility of the MVI, as determined by changes in 3-dimensional vestibulo-ocular reflex (3D VOR) gain and alignment compared to pre-intervention values and published data from subjects with normal vestibular function | Through study completion, an average of 1 year, that is: in visits 0, and 3 through 10
  3D VOR gain (eye velocity / -head velocity)
Assess the preliminary efficacy of the MVI, as determined by changes in 3-dimensional vestibulo-ocular reflex (3D VOR) gain and alignment compared to pre-intervention values and published data from subjects with normal vestibular function | Through study completion, an average of 1 year, that is: in visits 0, and 3 through 10
  3D VOR gain (eye velocity / -head velocity)
Assess the effects of MVI implantation on cochlear function, as indicated by changes in pure tone audiometry | through study completion, an average of 1 year, that is: in visits 0, and 3 through 10
  Pure tone audiometry (decibels [dB])
Assess the effects of MVI use on cochlear function, as indicated by changes in pure tone audiometry | through study completion, an average of 1 year, that is: in visits 0, and 3 through 10
  Pure tone audiometry (decibels [dB])
Assess the effects of MVI implantation on cochlear function, as indicated by changes in Consonant-vowel nucleus-consonant (CNC) speech recognition scores | through study completion, an average of 1 year, that is: in visits 0, and 3 through 10
  CNC speech recognition score (0-100% correct), higher scores means better outcome
Assess the effects of MVI use on cochlear function, as indicated by changes in Consonant-vowel nucleus-consonant (CNC) speech recognition scores | through study completion, an average of 1 year, that is: in visits 0, and 3 through 10
  CNC speech recognition score (0-100% correct), higher scores means better outcome
Assess the effects of MVI implantation on cochlear function, as indicated by changes in Arizona Biomedical (AzBio) sentence recognition scores | through study completion, an average of 1 year, that is: in visits 0, and 3 through 10
  AzBio sentence recognition score (0-100% correct), higher scores means better outcome
Assess the effects of MVI use on cochlear function, as indicated by changes in Arizona Biomedical (AzBio) sentence recognition scores | through study completion, an average of 1 year, that is: in visits 0, and 3 through 10
  AzBio sentence recognition score (0-100% correct), higher scores means better outcome

SECONDARY OUTCOMES:
Change in Vestibulo-ocular reflex (VOR) three-dimensional (3D) alignment to assess the preliminary efficacy of the MVI | In a period of up to 24 weeks, in visits 0, and 3 through 10
  Measured in degrees
Change in Ocular Vestibular Evoked Myogenic Potentials (oVEMP) to assess the effects of MVI implantation and use on utricular function | In a period of up to 24 weeks, in visits 0, and 3 through 10
  oVEMP peak-to-peak amplitude in microvolts
Change in Cervical Vestibular Evoked Myogenic Potentials (cVEMP) to assess the effects of MVI implantation and use on saccular function | In a period of up to 24 weeks, in visits 0, and 3 through 10
  cVEMP peak-to-peak amplitude in microvolts
Changes in utility scores on 36-Item Short Form Health Survey (SF-36) to assess the effects of MVI implantation and use on activities of daily living and quality of life | In a period of up to 24 weeks, in visits 0, 6, 8, and 10
  SF-36 Utility (No scale)
Changes in scores on Tinnitus Handicap Inventory (THI) to assess the effects of MVI implantation and use on activities of daily living and quality of life | In a period of up to 24 weeks, in visits 0, 6, 8, and 10
  THI score (0-100), higher scores means worse outcome
Changes in scores on Dizziness Handicap Inventory (DHI) to assess the effects of MVI implantation and use on activities of daily living and quality of life | In a period of up to 24 weeks, in visits 0, 6, 8, and 10
  DHI score (0-100), higher scores means worse outcome
Changes in scores on the Health Utilities Index 3 (HUI3) to assess the effects of MVI implantation and use on activities of daily living and quality of life | In a period of up to 24 weeks, in visits 0, 6, 8, and 10
  HUI3 scores (0-1), higher scores means better outcome
Changes in scores on the Vestibular Activities of Daily Living (VADL) to assess the effects of MVI implantation and use on activities of daily living and quality of life | In a period of up to 24 weeks, in visits 0, 6, 8, and 10
  VADL score (1-10), higher scores means worse outcome
Changes in scores on the Autophony Index (AI) to assess the effects of MVI implantation and use on activities of daily living and quality of life | In a period of up to 24 weeks, in visits 0, 6, 8, and 10
  AI score (0-104), higher scores means worse outcome
Changes in scores on the bilateral vestibular deficiency BVD-case definition subset of questions to assess the effects of MVI™ implantation and use on activities of daily living and quality of life | In a period of up to 24 weeks, in visits 0, 6, 8, and 10
  BVD-case definition subset of questions from the National Health Interview Survey 2008 Balance Questions (NHIS) score (no scale)
Change in Dynamic visual acuity (DVA) to assess the feasibility and preliminary efficacy of the MVI | In a period of up to 24 weeks, in visits 0 and 3 through 10
  DVA test score in log10 of the Minimum Angle Resolvable (LogMAR) units, as the difference between raw DVA LogMAR and static visual acuity LogMAR
Change in Bruininks-Oseretsky test of motor proficiency- balance subtest 2 (BOT2) score | In a period of up to 24 weeks, in visits 0, and 3 through 10
  BOT2 score (0-36), higher scores means better outcome
Change in Dynamic Gait Index (DGI) | In a period of up to 24 weeks, in visits 0, and 3 through 10
  DGI score (0-24), higher scores means better outcome
Change in gait characteristics using the GaitRite™ system | In a period of up to 24 weeks, in visits 0, and 3 through 10
  Gait speed analysis in meters per second

CONTACTS AND LOCATIONS:
Overall Officials: John P Carey MD (Independent/Nonconflicted IRB Protocol PI), Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
publication of de-identified data via peer-reviewed journals
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after publication and ending 36 months after publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal and signed data access agreement. Proposals should be directed to vestibularimplant@jhmi.edu.

REFERENCES:
- [Background] Sun DQ, Lehar M, Dai C, Swarthout L, Lauer AM, Carey JP, Mitchell DE, Cullen KE, Della Santina CC. Histopathologic Changes of the Inner ear in Rhesus Monkeys After Intratympanic Gentamicin Injection and Vestibular Prosthesis Electrode Array Implantation. J Assoc Res Otolaryngol. 2015 Jun;16(3):373-87. doi: 10.1007/s10162-015-0515-y. Epub 2015 Mar 20. PMID 25790951
- [Background] Sun DQ, Ward BK, Semenov YR, Carey JP, Della Santina CC. Bilateral Vestibular Deficiency: Quality of Life and Economic Implications. JAMA Otolaryngol Head Neck Surg. 2014 Jun;140(6):527-34. doi: 10.1001/jamaoto.2014.490. PMID 24763518
- [Background] Mitchell DE, Dai C, Rahman MA, Ahn JH, Della Santina CC, Cullen KE. Head movements evoked in alert rhesus monkey by vestibular prosthesis stimulation: implications for postural and gaze stabilization. PLoS One. 2013 Oct 17;8(10):e78767. doi: 10.1371/journal.pone.0078767. eCollection 2013. PMID 24147142
- [Background] Dai C, Fridman GY, Chiang B, Rahman MA, Ahn JH, Davidovics NS, Della Santina CC. Directional plasticity rapidly improves 3D vestibulo-ocular reflex alignment in monkeys using a multichannel vestibular prosthesis. J Assoc Res Otolaryngol. 2013 Dec;14(6):863-77. doi: 10.1007/s10162-013-0413-0. Epub 2013 Sep 8. PMID 24013822
- [Background] Ward BK, Agrawal Y, Hoffman HJ, Carey JP, Della Santina CC. Prevalence and impact of bilateral vestibular hypofunction: results from the 2008 US National Health Interview Survey. JAMA Otolaryngol Head Neck Surg. 2013 Aug 1;139(8):803-10. doi: 10.1001/jamaoto.2013.3913. PMID 23949355
- [Background] Valentin NS, Hageman KN, Dai C, Della Santina CC, Fridman GY. Development of a multichannel vestibular prosthesis prototype by modification of a commercially available cochlear implant. IEEE Trans Neural Syst Rehabil Eng. 2013 Sep;21(5):830-9. doi: 10.1109/TNSRE.2013.2259261. Epub 2013 May 1. PMID 23649285
- [Background] Davidovics NS, Rahman MA, Dai C, Ahn J, Fridman GY, Della Santina CC. Multichannel vestibular prosthesis employing modulation of pulse rate and current with alignment precompensation elicits improved VOR performance in monkeys. J Assoc Res Otolaryngol. 2013 Apr;14(2):233-48. doi: 10.1007/s10162-013-0370-7. Epub 2013 Jan 26. PMID 23355001
- [Background] Fridman GY, Della Santina CC. Progress toward development of a multichannel vestibular prosthesis for treatment of bilateral vestibular deficiency. Anat Rec (Hoboken). 2012 Nov;295(11):2010-29. doi: 10.1002/ar.22581. Epub 2012 Oct 8. PMID 23044664
- [Background] Rahman MA, Dai C, Fridman GY, Davidovics NS, Chiang B, Ahn J, Hayden R, Melvin TA, Sun DQ, Hedjoudje A, Della Santina CC. Restoring the 3D vestibulo-ocular reflex via electrical stimulation: the Johns Hopkins multichannel vestibular prosthesis project. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:3142-5. doi: 10.1109/IEMBS.2011.6090857. PMID 22255006
- [Background] Dai C, Fridman GY, Davidovics NS, Chiang B, Ahn JH, Della Santina CC. Restoration of 3D vestibular sensation in rhesus monkeys using a multichannel vestibular prosthesis. Hear Res. 2011 Nov;281(1-2):74-83. doi: 10.1016/j.heares.2011.08.008. Epub 2011 Aug 26. PMID 21888961
- [Background] Dai C, Fridman GY, Chiang B, Davidovics NS, Melvin TA, Cullen KE, Della Santina CC. Cross-axis adaptation improves 3D vestibulo-ocular reflex alignment during chronic stimulation via a head-mounted multichannel vestibular prosthesis. Exp Brain Res. 2011 May;210(3-4):595-606. doi: 10.1007/s00221-011-2591-5. Epub 2011 Mar 4. PMID 21374081
- [Background] Dai C, Fridman GY, Della Santina CC. Effects of vestibular prosthesis electrode implantation and stimulation on hearing in rhesus monkeys. Hear Res. 2011 Jul;277(1-2):204-10. doi: 10.1016/j.heares.2010.12.021. Epub 2010 Dec 31. PMID 21195755
- [Background] Della Santina CC. Regaining balance with bionic ears. Sci Am. 2010 Apr;302(4):68-71. doi: 10.1038/scientificamerican0410-68. No abstract available. PMID 20349578
- [Background] Fridman GY, Davidovics NS, Dai C, Migliaccio AA, Della Santina CC. Vestibulo-ocular reflex responses to a multichannel vestibular prosthesis incorporating a 3D coordinate transformation for correction of misalignment. J Assoc Res Otolaryngol. 2010 Sep;11(3):367-81. doi: 10.1007/s10162-010-0208-5. Epub 2010 Feb 23. PMID 20177732
- [Background] Della Santina CC, Migliaccio AA, Patel AH. A multichannel semicircular canal neural prosthesis using electrical stimulation to restore 3-d vestibular sensation. IEEE Trans Biomed Eng. 2007 Jun;54(6 Pt 1):1016-30. doi: 10.1109/TBME.2007.894629. PMID 17554821
- [Background] Hedjoudje A, Schoo DP, Ward BK, Carey JP, Della Santina CC, Pearl M. Vestibular Implant Imaging. AJNR Am J Neuroradiol. 2021 Jan;42(2):370-376. doi: 10.3174/ajnr.A6991. Epub 2020 Dec 24. PMID 33361382
- [Background] Chow MR, Ayiotis AI, Schoo DP, Gimmon Y, Lane KE, Morris BJ, Rahman MA, Valentin NS, Boutros PJ, Bowditch SP, Ward BK, Sun DQ, Trevino Guajardo C, Schubert MC, Carey JP, Della Santina CC. Posture, Gait, Quality of Life, and Hearing with a Vestibular Implant. N Engl J Med. 2021 Feb 11;384(6):521-532. doi: 10.1056/NEJMoa2020457. PMID 33567192
- [Result] Boutros PJ, Schoo DP, Rahman M, Valentin NS, Chow MR, Ayiotis AI, Morris BJ, Hofner A, Rascon AM, Marx A, Deas R, Fridman GY, Davidovics NS, Ward BK, Trevino C, Bowditch SP, Roberts DC, Lane KE, Gimmon Y, Schubert MC, Carey JP, Jaeger A, Della Santina CC. Continuous vestibular implant stimulation partially restores eye-stabilizing reflexes. JCI Insight. 2019 Nov 14;4(22):e128397. doi: 10.1172/jci.insight.128397. PMID 31723056
- [Derived] Schoo DP, Ayiotis AI, Fernandez Brillet C, Chow MR, Lane KE, Ward BK, Carey JP, Della Santina CC. Vestibular Implantation Can Work Even After More Than 20 Years of Bilateral Vestibular Hypofunction. Otol Neurotol. 2023 Feb 1;44(2):168-171. doi: 10.1097/MAO.0000000000003768. Epub 2022 Dec 17. PMID 36624598
- See also: Trial-related news updates and links to application — http://www.jhu.edu/vnel